CLINICAL TRIAL: NCT02588638
Title: Next Generation Sequencing Diagnostics - On the Road to Rapid Diagnostics for Rare Diseases
Acronym: NextGen-SE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ludger Schöls, Head of the Section Clinical Neurogenetics, University Hospital Tuebingen
Other Study IDs: NextGen-SE
Record Dates: First submitted 2015-10-15; First posted 2015-10-28 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Movement Disorder; Cognitive Decline
Keywords: NGS; Quality of life; Diagnosis; Rare disease; Next-generation sequencing
MeSH Terms: conditions — Movement Disorders; Cognitive Dysfunction; Disease; Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adult patients: Unclear movement disorder, unclear cognitive decline
- Patients < 18 years: Patients with (penetrating) suspected cerebral neurogenetic diseases

SUMMARY:
In the study, NextGen SE are on-hand a cohort comprising each 50 pediatric and 50 adult patients, and in which there are an unclear movement disorder or an unclear cognitive disorder, examines the following questions :

Primary:

* Number of diagnoses made by NGS

Secondary:

1. restriction of the quality of life by unclear disease
2. Cost of not purposeful preliminary diagnostics ( beyond the minimal diagnostic data set )
3. Impact of the diagnosis to therapy and follow-up examinations
4. Time to diagnosis

DETAILED DESCRIPTION:
In the study NextGen SE (single-center, prospective, open diagnostic study) are on-hand a cohort comprising each 50 pediatric and 50 adult patients, and in which there are an unclear movement disorder or an unclear cognitive disorder, examines the following questions:

Primary:

* Number of diagnoses made by next-generation sequencing (NGS)

Secondary:

1. Restriction of the quality of life by unclear disease
2. Cost of not purposeful preliminary diagnostics (beyond the minimal diagnostic data of the diagnosis to therapy and follow-up examinations
3. Time to diagnosis

ELIGIBILITY:
Inclusion Criteria:

For patients> 18 years

1. Unclear movement disorder

   o Progressive ataxia after minimal exclusion diagnostics: magnetic resonance tomography (MRT) (structural lesions such as cerebellar tumor, malformation) Laboratory (Vitamin B12, thyroid peroxidase (TPO) antibodies, glutamate decarboxylase (GAD) II-antibodies (AK) In medullary lesions: Liquor exclusion Friedreich ataxia (FRDA) and spinocerebellar ataxia type (SCA)1-2-3-6

   o Progressive para-spasticity by minimal exclusion diagnostics: MRT neuro axis (structural lesions such as cervical myelopathy) Laboratory (Vitamin B12, human T-cell lymphotrophic virus ((HTLV)-AK) In medullary lesions: Liquor
2. Unclear cognitive decline o After minimal exclusion diagnosis MRT (intracranial pressure, focal brain lesions explanatory) laboratory (Thyroid-stimulating hormone (TSH), TPO-AK, antibody profile limbic encephalitis) Liquor (inflammation, meningitis) Electroencephalography (EEG) (Status) Exclusion chromosome 9 open reading frame 72 (C9orf72)

For patients <18 years Patients with (penetrating) suspected cerebral neurogenetic diseases

* Unclear movement disorder (spasticity, ataxia, dyskinesia)
* Unclear cognitive disorder with probability of monogenic origin
* Fragile X Syndrome (Fra-X) at mentally retarded boy, Friedreich ataxia (FRDA) with ataxia should be genetically excluded

Exclusion Criteria:

For patients > 18 years

1. Lack of consent
2. symptom onset > 40 years of age
3. Sudden, abrupt beginning
4. As early as previous history of genetic diagnosis using next-generation sequencing (NGS), also in the form of a panel

For patients <18 years

1. injury brain disorders

   * On the basis of imaging
   * On the basis of medical history (premature baby, hypoxic-ischemic encephalopathy)
2. Inflammatory brain disorders

   * On the basis of imaging
   * On the basis of laboratory parameters (Oligoclonal fractions, cerebrospinal fluid (CSF) cell count increased)
3. Light, isolated mental developmental disorder or behavioral disorder (rare monogenetic) - (less than 2 standard deviartion of normal or - < 6 year olds - less than 1 year in development history back)
4. Sudden , abrupt beginning
5. Next-generation sequencing (NGS) also in the form of a panel

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unclear diagnoses
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of diagnoses made by next gereration sequency (NGS) | Within the study period of 18 months

SECONDARY OUTCOMES:
Restriction of the quality of life by unclear disease measured rated by Quality of Life Questionnaire (EQ5D), Depression Questionnaire (PHQ) | At day 1
  EQ-5D: Calculation preference value PHQ: Categorical analysis carried out by modified evaluation algorithms of the Diagnostic and Statistical Manual of Mental Disorders (DSM) -IV B
Cost of not purposeful preliminary diagnostics rated by questionnaire on costs (number of outpatient performances, stationary investigations, repetition 's imaging, genetic single diagnostics, high-priced diagnostic | At day 1
Time to diagnosis | At day 1
  For patients whose diagnosis can be made by NGS

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Schöls, Prof. Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital, Tübingen, Baden-Wurttemberg, Germany